CLINICAL TRIAL: NCT06601751
Title: Effects of Neurobic Exercise Program on Cognitive Abilities Among Older Adults With Mild Cognitive Impairment. A Randomised Controlled Trial.
Brief Title: Neurobic Exercise Program on Cognitive Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Memoona Awan
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive impairment; Neurobic exercise; Memory; ADL
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurobic exercise program (Experimental): Neurobic exercise program + Traditional Brain Exercises
  Interventions: Other: Neurobic Exercise Program
- Traditional brain exercises (Active Comparator): Traditional brain exercises calculation or memory games.
  Interventions: Other: Traditional Brain Exercise

INTERVENTIONS:
Other: Neurobic Exercise Program — 6 weeks to improve cognitive function, memory and overall brain health by introducing non-routine activities that require participants to utilise their multiple senses and remember sequences and patterns. Each activity would be performed 2-3 times/ session, for recalling the observation period set at 1 minute and at the end of the 9th week, the memory retention effect will be measured.
  Arms: Neurobic exercise program
Other: Traditional Brain Exercise — activities like calculation or memory games. These exercises will be conducted in 2 days/week for 60-minute sessions in 6 weeks. The memory retention effect will be measured at the end of the 9th week. It is intended to be the baseline for comparing the effectiveness of a neurobic exercise program.
  Arms: Traditional brain exercises

SUMMARY:
This research aims to investigate the significance of a neurobic exercise program on cognitive abilities, memory retention, activities of daily living (ADL), and quality of life (QOL) among older adults with mild cognitive impairment in Pakistan. It aims to find the long-term effects of a neurobic exercise program by comparing subjective and objective memory and its effects on quality of life.

DETAILED DESCRIPTION:
MCI is a condition marked by a noticeable decline in cognitive functions, it is often considered a precursor to more severe forms of dementia, making early intervention crucial. Neurobic exercises are designed to stimulate the brain through multiple senses and to create a novel thinking pattern. These exercises might include activities involving sight, smell, touch, taste, and hearing, structured over six weeks to challenge the brain with non-routine tasks that promote creative thinking and memory retention.

Neurobic exercise aims to maintain strength, flexibility, and mental health as you age.

However, most research has focused on older, healthy individuals or those with chronic conditions. Studies on elderly persons with MCI are rare, and there are limited studies on the long-term effects of improved memory function. This research aims to investigate the significance of a neurobic exercise program on cognitive abilities in older adults with mild cognitive impairment in Pakistan. It aims to find the long-term effects of a neurobic exercise program by comparing subjective and objective memory and its effects on quality of life. The findings will give insight to physiotherapists and multidisciplinary teams to improve memory retention, delay brain deterioration, and promote memory health and quality of life, making the intervention program a valuable guide.

ELIGIBILITY:
Inclusion Criteria:

* Older adults above 60
* Both male and female.
* Scored <24 on the Montreal Cognitive Assessment (MoCA).
* Scored >12 on the Modified Barthel ADL index (BAI).
* Ability to write and read as well as communicate well, willingness to participate in the study throughout the program

Exclusion Criteria:

* Neurological, musculoskeletal, psychiatric conditions, hearing loss and visual impairment.
* Older adults with a history of allergies to the food or flowers used in the activities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
MOCA (Montreal Cognitive Assessment) | 9 weeks
  The MOCA is a popular screening tool used to determine if cognitive impairment is present. It takes approximately ten minutes to complete. It evaluates visuospatial skills, attention, language, abstract reasoning, delayed recall, executive function, and orientation. MoCA is scored out of 30. A cut-off score of 26 signifies mild cognitive impairment.
Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | 9 weeks
  It is used to measure subjective memory. This test measures the informant's perception of the older person's cognitive decline. Older adults are required to compare their performance today with their performance ten years ago. Informants were asked to indicate the change on a 16-item scale from 1 (much improved) to 5 (much worse).
  The cut-off scores were based on the total score divided by the number of questions (average item score range 1- 5). Lower scores indicated better subjective memory performance.
Common Object Memory Test (COMT) | 9 weeks
  It is used to measure objective memory. The COMT was designed to assess age related memory impairments in individuals with various educational, language, and cultural backgrounds. It included repeated presentations of colour photographs containing 10 common objects (button, chair, clock, comb, cup, key, knife, leaf, scissors and umbrella) and multiple opportunities for participants to recall and recognise the original list. The total COMT scores were summed across these three steps, and the possible range was 0-90. Higher scores indicated better objective memory performance.

SECONDARY OUTCOMES:
Modified Barthel ADL Index (BAI) | 9 weeks
  The Barthel Index for Activities of Daily Living is an ordinal scale used to measure a person's ability to perform ten common daily activities, including feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfers (bed-to-chair), mobilityon level surfaces, and stair negotiation. A modified version by Collin and Wade uses a three-point scoring system (0 = unable, 1 = needs assistance, 2 = independent) with a total score ranging from 0 to 20. The assessment takes 2-5 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Aroosa Tariq, MS-NMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY ISLAMABAD
Locations (1):
- ZUK old home and health care center, Ghulam Haider Road, House# I-546-547, 342, 343, Faiz Building St#5, Committee Chowk, Rawalpindi., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No